CLINICAL TRIAL: NCT01672814
Title: A Randomized, Controlled Study of the Vedera™ KXS Microwave System With Corneal Collagen Cross-Linking Compared With Corneal Collagen Cross-Linking Alone for Eyes With Keratoconus
Brief Title: Microwave Treatment and Corneal Collagen Crosslinking for Keratoconus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cornea and Laser Eye Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VED-001
Record Dates: First submitted 2012-08-22; First posted 2012-08-27 (Estimated); Last update posted 2018-07-17 (Actual); Status verified 2018-07

CONDITIONS: Keratoconus
Keywords: Keratoconus; Collagen Crosslinking; Riboflavin; Microwave; Keraflex
MeSH Terms: conditions — Keratoconus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Keraflex combined with Crosslinking (Active Comparator): Vedera KXS microwave system used in conjunction with corneal collagen crosslinking performed with VibeX (Riboflavin ophthalmic solution)and the KXL UV System
  Interventions: Drug: riboflavin ophthalmic solution; Device: Vedera KXS Microwave System
- Corneal collagen crosslinking alone (Active Comparator): Corneal collagen crosslinking alone performed with VibeX (Riboflavin Ophthalmic Solution)and the KXL UV system
  Interventions: Drug: riboflavin ophthalmic solution

INTERVENTIONS:
Drug: riboflavin ophthalmic solution — Administration of riboflavin every 2 minutes for 20 minutes
  Other Names: VibeX
Device: Vedera KXS Microwave System — The Vedera KXS dose will be based on the pre-treatment manifest refraction spherical equivalent (MRSE), to be administered one day prior to the CXL procedure.
  Other Names: Keraflex
  Arms: Keraflex combined with Crosslinking

SUMMARY:
This study compares the outcomes of the Vedera KXS procedure (a microwave-based procedure, also known as Keraflex) combined with corneal collagen crosslinking to corneal collagen crosslinking alone for the treatment of keratoconus. The goal is to improve corneal shape in patients with keratoconus.

DETAILED DESCRIPTION:
The objective of this study is to compare the safety and efficacy of the Vedera KXS (a microwave-based procedure) combined with corneal collagen cross-linking performed with VibeX (Riboflavin Ophthalmic Solution)and the KXL System to corneal collagen cross-linking alone in reducing corneal curvature in patients with keratoconus. Patients will be randomized into one of two treatment groups: Vedera KXS combined with corneal collagen cross-linking or collagen cross-linking alone. The Vedera KXS procedure performs a controlled application of microwave energy in an annular configuration. The goal of this procedure is to reshape the cornea to flatten the cornea and improve corneal topography in patients with keratoconus. The primary goal of collagen crosslinking is to stabilize the corneal shape in keratoconus and prevent progression of the disease. Moreover, investigations of crosslinking have shown the procedure not only to decrease keratoconus progression, but also to decrease the steepness of the cone and improve uncorrected and best corrected visual acuity in some cases. Since the mechanism of improvement differs between the procedures, this study will compare the combined microwave/crosslinking treatment to crosslinking alone.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 18 years of age
* Provide written consent and sign a HIPAA form
* Willingness and ability to follow all instructions and comply with schedule for follow-up visits
* For females capable of becoming pregnant, agree to have urine pregnancy testing performed prior to treatment; must not be lactating, and must agree to use a medically acceptable form of birth control for at least one week prior to the treatment and continue to use the method until 1 month after the last dose of investigational product.
* Having topographic evidence of keratoconus which is graded as moderate or severe keratoconus
* Presence of central or inferior steepening on the Pentacam map
* Steepest keratometry (Kmax) value greater than or equal to 51.00D
* BSCVA of 80 letters or fewer for keratoconus on ETDRS chart
* Contact lens wearers only: remove contact lenses one week prior to the screening refraction
* Contact lens wearers only: manifest refraction must be stable between two visits that occur at least 7 days apart.

Exclusion Criteria:

* Contraindications, sensitivity or known allergy to the use of the test articles(S) or their components
* If female, be pregnant, nursing, or planning a pregnancy or have a positive urine pregnancy test at Visit 2 prior to treatment or during the course of the study
* Eyes classified as either normal,atypical normal,keratoconus suspect or mild keratoconus on the severity grading scheme
* A history of the insertion of INTACS in the eye to be treated
* A history of previous limbal relaxing incision procedure in the eye to be treated
* Corneal pachymetry that is <350 microns at the thinnest point measured by Pentacam in the eye to be treated
* Eyes which are aphakic
* Eyes which are pseudophakic and do not have a UV blocking lens implanted
* Previous ocular condition (other than refractive error) in the eye to be treated that may predispose the eye for future complications.
* A history of delayed epithelial healing in the eye to be treated
* Patients with nystagmus or any other condition that would prevent a steady gaze during the treatment or other diagnostic tests
* Patients with a current condition that, in the investigator's opinion,would interfere with or prolong epithelial healing
* Taking Vitamin C (ascorbic acid) supplements within 1 week of the cross-linking treatment
* A history of previous corneal cross-linking treatment in the eye to be treated
* Have used an investigational drug or device within 30 days of the study or be concurrently enrolled in another investigational drug or device study within 30 days of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2012-08; Primary Completion 2017-06-01 (Actual); Study Completion 2017-06-01 (Actual)

PRIMARY OUTCOMES:
Maximum Keratometry | 12 months
  The change in maximum keratometry (Kmax) from baseline will be evaluated at 12 months for all eyes randomized to the two treatment groups. As a secondary analysis of this endpoint,the change in maximum keratometry (Kmax)from baseline will be evaluated at 1,3 and 6 months for all eyes.

SECONDARY OUTCOMES:
Manifest refraction | 12 months
  The change in manifest refraction spherical equivalent from baseline will be evaluated at 12 months. As secondary analysis of this endpoint, a repeated measures analysis of variance will be conducted to assess the profile of the treatments across time at 1,3,and 6 months to look at the effect of wound healing on this variable.

OTHER OUTCOMES:
Visual Acuity | 12 months
  Change in BSCVA (best spectacle corrected visual acuity) and UCVA (uncorrected visual acuity) compared to the baseline examination will be evaluated at 12 months postoperatively. As a secondary analysis of this endpoint, data across time from 1,3, and 6 months following the procedure will be analyzed.
Endothelial cell density | 12 months
  Endothelial cell count will be obtained using specular microscopy (Konan Medical) prior to KXS/CXL and CXL alone treatment and at 12 months postoperatively.

CONTACTS AND LOCATIONS:
Overall Officials: Peter S Hersh, MD, Principal Investigator — Cornea and Laser Eye Institute
Locations (1):
- Cornea and Laser Eye Institue - Hersh Vision Group, Teaneck, New Jersey, United States